CLINICAL TRIAL: NCT06208176
Title: Targeting Multimodal Hallucinations With fMRI-guided High-definition Transcranial Direct Current Stimulation (HD-tDCS) in Schizophrenia
Brief Title: HD-tDCS for Hallucinations
Acronym: TARGET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-A01629-36
Record Dates: First submitted 2023-12-12; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia; Hallucinations
Keywords: schizophrenia; non-invasive brain stimulation; fMRI; HD-tDCS; hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Intervention Model Description: The study is a multicentre, prospective, randomised, double-blind, parallel group, sham-controlled, two-arm clinical trial. Arm one is repeated active HD-tDCS guided by the fMRI-capture of hallucinations. Arm two is the blinded repeated sham HD-tDCS guided by the fMRI-capture of hallucinations
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients and experimenters (including tDCS operator) will not be informed about the nature (active or sham) of the stimulation they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulation group (Active Comparator): 23 patients will receive 20 sessions of active HD-tDCS
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), active condition
- placebo stimulation group (Placebo Comparator): High-definition transcranial direct current (HD-tDCS), sham condition
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), sham condition

INTERVENTIONS:
Procedure: High-definition transcranial direct current (HD-tDCS), active condition — Patients will receive 20 sessions of active HD-tDCS for a duration of 20min. Sessions will be delivered twice-daily over 2 weeks on the 5 consecutive working days. The number of electrodes used, electrode placement on the scalp (based on EEG 10/10), and the individual currents that need to be injected from each electrode will be determined based on the brain networks identified as involved in their hallucinations during a fMRI acquisition performed at baseline, and computed using a neurotargeting software that allows determining optimal electrode montages for achieving maximal brain current flow in the targeted brain region.
  Arms: active stimulation group
Procedure: High-definition transcranial direct current (HD-tDCS), sham condition — Participants will receive 20 sessions of sham HD-tDCS, which will be delivered following the same procedures as active HD-tDCS. However, stimulation will only be administered in the initial 30 seconds of the 20-minute period, with no further stimulation during the remaining duration. This approach aims to replicate the tingling sensation commonly associated with active stimulation.
  Arms: placebo stimulation group

SUMMARY:
One in three patients with schizophrenia experiences hallucinations that are refractory to conventional pharmacotherapy. For refractory auditory hallucinations, transcranial direct current stimulation -tDCS- has been proposed as a novel therapeutic approach. Although promising beneficial effects on auditory hallucinations have been found by targeting the left frontal and temporoparietal cortex, the high variability observed in clinical response leaves much room for optimizing stimulation parameters. For instance, options should go beyond the left temporoparietal junction as a unique and single target of hallucinations, taking into account the personalization of the targeting based on the actual brain networks involved in hallucinations, including those beyond the auditory modality, as well as multimodal hallucinations.

The present study will take advantage of recent technological developments to propose a personalized therapeutic strategy to alleviate hallucinations in schizophrenia. This will involve:

* the simultaneous targeting of multiple brain regions with High-Definition (HD)-tDCS, which is known for its precise and longer-lasting effects compared to conventional tDCS.
* and the fMRI-capture of hallucinations, using a precise and reliable data-driven approach to identify the functional brain networks recruited during hallucinations.

The aim of the study is to assess whether repeated sessions of HD-tDCS guided using the fMRI capture of hallucinations can reduce multimodal hallucinations in patients with schizophrenia, compared to sham sessions of HD-tDCS.

DETAILED DESCRIPTION:
The study is a multicentre, prospective, randomised, double-blind, parallel group, sham-controlled, two-arm clinical trial. Arm one is repeated active HD-tDCS guided using the fMRI-capture of hallucinations (20 sessions of stimulation over 10 days, 20 min/session). Arm two is the blinded sham repeated HD-tDCS guided by the fMRI-capture of hallucinations (20 sessions of sham stimulation over 10 days, 20 min/session).

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged between 18 and 50
* Diagnosis of schizophrenia according to DSM 5.0 criteria
* Presence of dailyfrequent hallucinations (> 2 / hour) despite the optimization of the antipsychotic dosage and molecule (based on the prescriber's judgment) for at least 6 weeks. The presence of such daily frequent refractory hallucinations will be operationalized by an interview with a trained psychiatrist.
* Patient under curatorship/guardianship or not
* Covered by a public health insurance
* Understanding French language
* Signed written informed consent after being informed about the study

Exclusion Criteria:

* Other disabling Axis Inpsychiatric conditions including a current diagnosis of a major depressive episode (uni- or bi- polar disorder) according to DSM 5, and substance use disorder (except tobacco)
* Use of hallucinogenic drugs
* Contraindications for magnetic resonance imaging or tDCS (neurologic stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid derivation, metallic splinters in the eyes, cochlear implants, severe claustrophobia)
* Changes in the total PSAS and PANSS score of at least 15% between screening/inclusion (T0) and baseline visits (T1). This criterion will ensure the stability of symptoms before treatment.
* Pregnancy (controlled by urine pregnancy test in women of childbearing potential) or breastfeeding
* A clinical condition requiring inpatient procedure under constraint

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in hallucinations | 6 months
  Comparison between the active HD-tDCS group and the sham HD-tDCS group of the change in multimodal hallucinations between baseline (V1, within 1 week before the first HD-tDCS session) and after the 20 HD-tDCS sessions (V2, within 1 week of the last HD-tDCS session). Change in hallucinations will be measured as the percentage change in score on the Psychosensory Hallucination Scale

SECONDARY OUTCOMES:
Long-term changes in hallucinations | 6 months
  Comparisons between active and sham HD-tDCS groups of the change in multimodal hallucinations (assessed with the PSAS, in percent) between baseline and follow-up assessments at one month and three months after the 20 sessions of HD-tDCS.
Change in symptoms of schizophrenia | 6 months
  Comparisons between active and sham HD-tDCS groups of the change in other symptoms of schizophrenia between baseline (V1, within 1 week before first stimulation) and post-intervention (V2, within 1 week after last stimulation), and follow-up assessments (V3: at one month, V4: at 3 months). Symptoms of schizophrenia will be measured by the total score at the Positive and Negative Syndrome Scale - PANSS , and by the scores in the five subdimensions of the PANSS (positive, negative, depression, disorganization, and grandiosity/excitement).
Change in social functioning | 6 months
  Comparisons between active and sham HD-tDCS groups of change in social functioning measured by the Social and Occupational Functioning Assessment Scale - SOFAS (Goldman et al., 1992) between baseline (V1, within 1 week before first stimulation) and follow-up assessments, one month (V3) and three months (V4) after the intervention
Changes in source-monitoring performance | 6 months
  Source monitoring performance will be evaluated using a specific source monitoring task. Source-monitoring accuracy scores (range 0-100) will be calculated as proportions of accurate source attributions for each source
Changes in brain connectivity | 6 months
  Comparisons between active and sham HD-tDCS groups of changes in brain connectivity within the hallucination-related network, measured with fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided